CLINICAL TRIAL: NCT00032123
Title: A Phase II Study Of OSI-774 (NSC 718781) In Unresectable Or Metastatic Adenocarcinoma Of The Stomach And Gastroesophageal Junction
Brief Title: Erlotinib in Treating Patients With Locally Advanced or Metastatic Stomach Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069259; SWOG-S0127
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; stage IV esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus; recurrent esophageal cancer; recurrent gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor.

PURPOSE: Phase II trial to study the effectiveness of erlotinib in treating patients who have locally advanced or metastatic stomach cancer or cancer of the gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate of patients with locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction treated with erlotinib. (Gastric stratum temporarily closed to accrual as of 03/01/2003.)
* Determine the frequency and severity of toxic effects of this drug in these patients.
* Determine the overall survival and time to treatment failure in patients treated with this drug.
* Determine the value of intratumoral expression of epidermal growth factor receptor in predicting patient response to this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to cancer site (stomach vs gastroesophageal junction). (The gastric stratum is temporarily closed to accrual as of 03-01-2003.)

Patients receive oral erlotinib once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 40-80 patients (20-40 per stratum) will be accrued for this study within 14-40 months. (The gastric stratum is temporarily closed to accrual as of 03-01-2003.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the stomach* or gastroesophageal (GE) junction

  * GE junction tumors include esophageal tumors arising 5 cm from the anatomic GE junction or in the gastric cardia
  * Locally advanced (i.e., unresectable) or metastatic disease NOTE: *Gastric stratum temporarily closed to accrual as of 03/01/2003
* Unidimensionally measurable disease

  * Target lesion must not be in previously irradiated field unless there is documentation of clear progression
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 1.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No recent myocardial infarction
* No unstable angina
* No life-threatening arrhythmia

Gastrointestinal:

* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No active peptic ulcer disease
* Must be able to swallow and/or receive enteral medications via gastrostomy feeding tube
* No intractable nausea or vomiting

Ophthalmic:

* No history of corneal disease, including:

  * Dry eye syndrome or Sjögren's syndrome
  * Keratoconjunctivitis sicca
  * Exposure keratopathy
  * Fuch's dystrophy
  * Other active disorders of the cornea

Other:

* HIV negative
* No active or uncontrolled infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* No severe psychiatric disorders
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy
* No concurrent anticancer immunotherapy

Chemotherapy:

* No prior chemotherapy for advanced or metastatic gastric cancer
* At least 8 weeks since prior adjuvant chemotherapy or chemotherapy given as a radiosensitizer and recovered
* No concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery:

* At least 4 weeks since prior surgical procedure for stomach* or GE cancer and recovered
* No prior surgical procedures that would affect absorption NOTE: *Gastric stratum temporarily closed to accrual as of 03/01/2003

Other:

* No prior investigational drugs
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-06; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Dragovich, MD, PhD, Study Chair — University of Arizona
Locations (107):
- United States (106):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Western New York Urology Associates, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at the University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Dragovich T, McCoy S, Fenoglio-Preiser CM, Wang J, Benedetti JK, Baker AF, Hackett CB, Urba SG, Zaner KS, Blanke CD, Abbruzzese JL. Phase II trial of erlotinib in gastroesophageal junction and gastric adenocarcinomas: SWOG 0127. J Clin Oncol. 2006 Oct 20;24(30):4922-7. doi: 10.1200/JCO.2006.07.1316. PMID 17050876
- [Result] Dragovich T, McCoy S, Urba SG, et al.: SWOG 0127: phase II trial of erlotinib in GEJ and gastric adenocarcinomas. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-49, 2005.